CLINICAL TRIAL: NCT00155129
Title: The Role of Calcitonin Gene-Related Peptide(CGRP)and Nociceptin in the Pathogenesis of Migraine
Brief Title: The Role of CGRPand Nociceptin in Migraine
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: National Taiwan University Hospital (Other)
Other Study IDs: 9361701099; 9361701099
Record Dates: First submitted 2005-09-09; First posted 2005-09-12 (Estimated); Last update posted 2005-09-12 (Estimated); Status verified 2005-06

CONDITIONS: Migraine; Headache
Keywords: migraine; CGRP; nociceptin
MeSH Terms: conditions — Migraine Disorders; Headache

STUDY DESIGN:
Observational Model: Defined Population | Time Perspective: Other

SUMMARY:
The release of the neuropeptide calcitonin gene-related peptide (CGRP) is thought to play a causative role in migraine. Nociceptin immunoreactivity and ORL-1 mRNA have been detected in human trigeminal ganglia where it was co-localized with CGRP. It may play a role in migraine pathogenesis. We are collecting the blood samples of migraineurs for analysis of these neuropeptides.

DETAILED DESCRIPTION:
The release of the neuropeptide calcitonin gene-related peptide (CGRP) is thought to play a causative role in migraine. Nociceptin immunoreactivity and ORL-1 mRNA have been detected in human trigeminal ganglia where it was co-localized with CGRP. It may play a role in migraine pathogenesis. We are collecting the blood samples of migraineurs for analysis of these neuropeptides.

ELIGIBILITY:
Inclusion Criteria: patients with headache -

Exclusion Criteria: fever, congenital anomaly, CNS organic lesions

-

Ages: 3 Years to 50 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Child, Adult
Enrollment: 200
Dates: Start 2005-01; Study Completion 2005-06

CONTACTS AND LOCATIONS:
Overall Officials: Pi-Chuan Fan, Principal Investigator — Department of Pediatric, NTUH
Locations (1):
- Department of Pediatrics, Taipei, Taiwan